CLINICAL TRIAL: NCT06263504
Title: The Influence of Complex Correction of Dental and Musculoskeletal Systems on the Frequency of Relapses of Functional Disorders in Patients With Dental Pathologies: a Randomized Pilot Clinical Trial
Brief Title: The Influence of Complex Correction of Dental and Musculoskeletal Systems on the Frequency of Relapses of Functional Disorders in Patients With Dental Pathologies.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NMSI DENTMASTER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM001
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Malocclusion; Musculoskeletal Disorder
Keywords: Malocclusion; Musculoskeletal Disorders; orthodontics; dental prosthetics; complex correction of the dental system
MeSH Terms: conditions — Malocclusion; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- receive standard treatment group (Active Comparator)
  Interventions: Procedure: at correcting malocclusions or restoring the integrity of the dentition
- comprehensive treatment group (Experimental)
  Interventions: Procedure: comprehensive treatment, including not only dental correction of bite or restoration of the integrity of the dentition, but also correction of disorders of the musculoskeletal system.

INTERVENTIONS:
Procedure: at correcting malocclusions or restoring the integrity of the dentition — Patients in this group will receive standard treatment aimed solely at correcting malocclusions or restoring the integrity of the dentition without interfering with the musculoskeletal system.
  Arms: receive standard treatment group
Procedure: comprehensive treatment, including not only dental correction of bite or restoration of the integrity of the dentition, but also correction of disorders of the musculoskeletal system. — ): Patients will receive comprehensive treatment, including not only dental correction of bite or restoration of the integrity of the dentition, but also correction of disorders of the musculoskeletal system.
  Arms: comprehensive treatment group

SUMMARY:
In influence of complex correction of dental and musculoskeletal systems on the frequency of relapses of functional disorders in patients with somatic pathologies: a randomized pilot study there will be two groups: Group 1 (control group): Patients in this group will receive standard treatment aimed solely at correcting malocclusions or restoring the integrity of the dentition without interfering with the musculoskeletal system.

Group 2 (experimental group): Patients will receive comprehensive treatment, including not only dental correction of bite or restoration of the integrity of the dentition, but also correction of disorders of the musculoskeletal system.

The endpoints will be :

Primary endpoint:

• Frequency of relapses and repeated requests for correction of disorders bite or restoration of the integrity of the dentition within 12 months after treatment.

Secondary endpoints:

* Change in pain intensity measured by visual analog scale (VAS).
* Improvement of functional indicators of the temporomandibular joint, including range of motion.
* Improved quality of life, assessed using the OHRQoL (Oral Health Related Quality) scale All endpoints will be evaluated within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed malocclusion or dentition insufficiency, confirmed by a dentist.

  * Presence of diseases of the musculoskeletal system, confirmed orthopedist or rheumatologist.
  * Acquired limb deformities (for example, flat feet, valgus or varus deformity).
  * Deforming dorsopathies (kyphosis, lordosis, scoliosis, osteochondrosis).
  * Consent to participate in the study and follow the treatment protocol.
  * Sufficient general physical and mental fitness to participate in the study

Exclusion Criteria:

* Systemic diseases affecting bone metabolism (eg osteoporosis).

  * Progressive neurological diseases.
  * Current treatment with steroids or immunosuppressive drugs.
  * Presence of malignant neoplasms.
  * Psychiatric disorders that prevent compliance protocol.
  * Pregnancy or lactation period.
  * Carrying out dental or orthopedic treatment in recent 6 months.
  * Skeletal malocclusions.
  * Diseases of the temporomandibular joint.
  * Congenital pathologies of the musculoskeletal system.
  * Arthropathy.
  * Systemic connective tissue diseases.
  * Biomechanical lesions of the musculoskeletal system.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of relapses and repeated requests for correction of disorders bite or restoration of the integrity of the dentition. | 12 months

SECONDARY OUTCOMES:
Change in pain intensity measured by visual analog scale (VAS). | 12 months
  A Visual Analogue Scale - VAS Purpose: pain intensity assessments
  Interpretation:
  0 points - no violations; 1-3 points - mild pain (mild impairment); 4-6 points - moderate pain (moderate impairment); 7-8 points - severe pain (severe impairment); 9-10 points - unbearable pain (absolute violations).
Changes in functional parameters of the temporomandibular joint, including range of motion. joint, including range of motion. | 12 month
  0- No changes
  1. The changes are positive
  2. Changes are negative
Improved quality of life, assessed using the OHRQoL (Oral Health Related Quality) scale | 12 month
  Change in quality of life, assessed by the OHRQoL-Oral Health Related Quality of Life scale. Index of the impact of oral health on quality of life (OHIP - Oral Health Impact Profile).
  The Oral Health Impact Index (OHIP) includes 49 questions covering 7 dimensions: functional limitation, physical pain, psychological discomfort, physical, psychological, social discomfort and lack of confidence. Scores for each question range from 0 (never) to 4 (always), meaning the maximum possible total score is 196. The minimum score, 0, indicates no impact of oral health problems on quality of life. The higher the score, the greater the impact on quality of life the patient experiences

CONTACTS AND LOCATIONS:
Locations (1):
- Nmsi Dentmaster, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided